CLINICAL TRIAL: NCT03920085
Title: Clinical Evaluation of LifeScan Blood Glucose Monitoring Systems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LifeScan Scotland Ltd (Industry)
Collaborators: MAC Clinical Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 3177234
Record Dates: First submitted 2019-04-05; First posted 2019-04-18 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2019-03

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- LifeScan BGMSs (Experimental): OneTouch Verio, OneTouch Select Plus and OneTouch Ultra Blood Glucose Monitoring Systems (BGMSs) tested using subject capillary blood and compared to a reference instrument (YSI 2900).
  Interventions: Device: OneTouch Verio; Device: OneTouch Select Plus; Device: OneTouch Ultra

INTERVENTIONS:
Device: OneTouch Verio — OneTouch Verio Blood Glucose Monitoring System.
Device: OneTouch Select Plus — OneTouch Select Plus Blood Glucose Monitoring System.
Device: OneTouch Ultra — OneTouch Ultra Blood Glucose Monitoring System.

SUMMARY:
Study to determine the performance of the LifeScan BGMS when conducted at MAC clinical site.

DETAILED DESCRIPTION:
This study will evaluate the performance of the MAC clinical site to evaluate accuracy performance of LifeScan blood glucose monitoring systems as it is conducted at other LifeScan UK affiliated clinic sites. Multiple LifeScan Blood Glucose Monitoring System (BGMS) will be tested with production lots which have passed release testing.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be enrolled in LifeScan Patient Registry.
* Participants must have read the Information sheet and signed an informedconsent form >prior to study participation.
* Participants must be 16 years or older.
* Participants must be diagnosed with Diabetes

Exclusion Criteria:

> Participants not enrolled in the LifeScan Patient Registry

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2019-02-05 (Actual); Study Completion 2019-02-05 (Actual)

PRIMARY OUTCOMES:
Clinical Evaluation of Blood Glucose result (mg/dl) from LifeScan Blood Glucose Monitoring Systems by comparison of a blood glucose result (mg/dl) obtained from a reference instrument (YSI2900) to demonstrate accuracy (%). | Less than 30 minutes
  Clinical Evaluation of Blood Glucose result (mg/dl) from LifeScan Blood Glucose Monitoring Systems by comparison of a blood glucose result (mg/dl) obtained from a reference instrument (YSI2900) to demonstrate accuracy (%).

CONTACTS AND LOCATIONS:
Locations (1):
- MAC Clinical Research, Manchester, United Kingdom